CLINICAL TRIAL: NCT06984276
Title: Efficacy Of Ultrasound Guided Bilateral Pectoral Nerve Block Versus Bilateral Transverse Thoracic Plane Block In Pediatric Patients Undergoing Corrective Cardiac Surgeries Requiring Cardiopulmonary Bypass Via Median Sternotomy: A Randomized Controlled Trial.
Brief Title: Ultrasound Guided Bilateral Pectoral Nerve Block Versus Bilateral Transverse Thoracic Plane Block In Pediatric Patients Undergoing Corrective Cardiac Surgeries Requiring Cardiopulmonary Bypass Via Median Sternotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Mahmoud Elfiky, Assistant Lecturer of Anesthesia, Surgical ICU and Pain Management, Cairo University Hospitals., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-263-2024
Record Dates: First submitted 2025-05-20; First posted 2025-05-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Ultrasound; Pectoral Nerve Block; Transverse Thoracic Plane Block; Pediatric Patients; Corrective Cardiac Surgeries; Cardiopulmonary Bypass; Median Sternotomy
MeSH Terms: interventions — Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients will receive o.5 ug/kg/hr fentanyl infusion all through the whole operation.
  Interventions: Drug: Control
- Pectoral nerves group (Experimental): This group will receive fentanyl infusion at a dose of (0.5 μg/kg/hr) all through the whole operation, plus ultrasound guided bilateral pectoral nerves (PECS) Block which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .
  Interventions: Other: Pectoral nerves (PECS)
- Transversus thoracic muscle plane block group (Experimental): This group will receive fentanyl infusion at a dose of (0.5 μg/kg/hr) all through the whole operation, plus Ultrasound guided bilateral transversus thoracic muscle plane block (TTPB) which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .
  Interventions: Other: Transversus thoracic muscle plane block (TTPB)

INTERVENTIONS:
Drug: Control — Patients will receive o.5 ug/kg/hr fentanyl infusion all through the whole operation.
  Other Names: Fentanyl
  Arms: Control group
Other: Pectoral nerves (PECS) — This group will receive fentanyl infusion at a dose of (0.5 μg/kg/hr) all through the whole operation, plus ultrasound guided bilateral pectoral nerves (PECS) Block which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .
  Other Names: Bupivacaine 0.25% and lidocaine 1%
  Arms: Pectoral nerves group
Other: Transversus thoracic muscle plane block (TTPB) — This group will receive fentanyl infusion at a dose of (0.5 μg/kg/hr) all through the whole operation, plus Ultrasound guided bilateral transversus thoracic muscle plane block (TTPB) which will be done by injecting 0.4 ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .
  Other Names: Bupivacaine 0.25% and lidocaine 1%)
  Arms: Transversus thoracic muscle plane block group

SUMMARY:
This randomized, double-blinded, study aims to compare the efficacy of intraoperative and postoperative pain control while using bilateral ultrasound guided the pectoral nerves (PECS) versus transversus thoracic muscle plane block (TTPB) in pediatric patients undergoing corrective cardiac surgeries.

DETAILED DESCRIPTION:
Good perioperative analgesia in cardiac surgical patients helps early recovery, ambulation, and early discharge from the Intensive Care Unit (ICU). Traditional use of nonsteroidal anti-inflammatory drugs (NSAIDs) and opioids associated with adverse effect commonly used for pain control postoperative.

The transversus thoracic muscle plane block (TTPB) is a recently advised regional anesthesia method that provides analgesia to the anterior chest wall and was initially introduced by Ueshima et al. in 2015 .

The pectoral nerves (PECS) block has evolved to be two different types: PECS I and PECS II. In PECS I block, anesthetic is injected in the interfacial plane between the pectoralis major and minor muscles at the 3rd rib, blocking the lateral and medial pectoral nerves. The PECS II block, which was also developed by Blanco in 2012.

The PECS block has been well established for its use in breast surgery for the adult population. , However, there has been a recent push in the last couple of years to find more about other uses for these types of blocks, especially in cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months - 7 years.
* Gender: both sexs .
* Risk Adjustment for Congenital Heart Surgery (RACHS) II and III.
* Patients undergoing cardiac surgeries requiring cardiopulmonary bypass with midline sternotomy incision.

Exclusion Criteria:

* Patients whose parents or legal guardians refuse to participate.
* Preoperative mechanical ventilation.
* Patients in coma, mental retardation, neurological disease, or on drugs affecting the behaviour.
* Preoperative inotropic drug infusion.
* (Bleeding disorders (drug induced i.e., coumadin; or genetic e.g. hemophilia; or acquired e.g. disseminated intravascular coagulation [DIC]), coagulopathy: Partial Thromboplastin Time (PTT) > 40 seconds, International Normalized Ratio (INR) > 1.4, platelet count < 100x10⁹.
* Known or suspected allergy to any of the studied drugs.
* Severe pulmonary hypertension (mean resting blood pressure in pulmonary arteries is above 70mmHg).
* Cardiopulmonary bypass time more than 90 minutes.
* local infection.
* Significant Renal impairment (creatinine more than 1.2mg/dl)
* Aortic cross-clamp time more than 45 minutes.
* Total time from induction till intensive Care Unit (ICU) transfer more than 4 hours and 30 mins.

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The total dose of intraoperative fentanyl | Intraoperatively
  The total dose of intraoperative fentanyl will be recorded

SECONDARY OUTCOMES:
Degree of pain | 12 hours postoperatively
  Pain will be assessed by the pediatric observational 10-point scale "Face, Leg, Activity, Cry, Consolability (FLACC) pain score immediately after admission to intensive care unit (ICU) then at 60 min, 2 hours, 4hours, 8hours and 12 hours postoperatively.
  If the patient FLACC score equal or more than 4, patient will receive Fentanyl I.V 1 mic /kg .
Heart rate | 12 hours postoperatively
  Heart rate (HR) immediately after admission to Intensive Care Unit (ICU) then at 60 min, 2 hours, 4hours, 8 hours and 12 hours
Mean arterial pressure | 12 hours postoperatively
  Mean arterial pressure (MAP) immediately after admission to Intensive Care Unit (ICU) then at 60 min, 2 hours, 4hours, 8 hours and 12 hours
Total consumption of Fentanyl | 12 hours postoperatively
  Total consumption of Fentanyl during the 1st 12 hours postoperatively will be recorded
Time to 1st rescue analgesia | 12 hours postoperatively
  Time to 1st rescue analgesia post operatively which will be defined to be the elapsed time between giving the block and a patient FLACC score equal or more than 4.
Time of Extubation | 12 hours postoperatively
  Time of Extubation will be recorded
The incidence of opioid complications | 12 hours postoperatively
  The incidence of opioid complications like postoperative nausea and vomiting (PONV), hematoma formation, itching will be recorded
The incidence of Local anatectic toxicity | 12 hours postoperatively
  The incidence of Local anatectic toxicity like neurologic symptoms (seizures, and ultimately neurologic depression with respiratory arrest, coma, or both) and Cardiovascular symptoms may include an hypertensive , tachycardia, cardiac depression with bradycardia, myocardial depression, conduction block, asystole, and cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year
Supporting Information: Study Protocol
Time Frame: After the end of study for one year
Access Criteria: The data will be available upon a reasonable request from the corresponding author